CLINICAL TRIAL: NCT01767116
Title: A Randomized, Double-blind, Controlled Study to Evaluate the Efficacy and Safety of the Combination of ABT-450/Ritonavir/ABT-267 (ABT-450/r/ABT-267) and ABT-333 With and Without Ribavirin (RBV) in Treatment-Naive Adults With Genotype 1b Chronic Hepatitis C Virus (HCV) Infection (PEARL-III)
Brief Title: A Study to Evaluate Chronic Hepatitis C Infection in Adults With Genotype 1b Infection
Acronym: PEARL-III
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AbbVie (prior sponsor, Abbott) (Industry)
Responsible Party: Sponsor
Organization: AbbVie (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: M13-961; 2012-003687-52 (EudraCT Number)
Record Dates: First submitted 2012-11-30; First posted 2013-01-14 (Estimated); Results first posted 2015-01-06 (Estimated); Last update posted 2021-07-12 (Actual); Status verified 2021-07

CONDITIONS: Chronic Hepatitis C Infection
Keywords: Interferon-Free; Hepatitis C Genotype 1b; Chronic Hepatitis C; Hepatitis C Virus; Hepatitis C; Treatment-Naive; Paritaprevir; Ombitasvir; Dasabuvir; Viekira PAK; Ribavirin
MeSH Terms: conditions — Hepatitis C, Chronic; Hepatitis C | interventions — dasabuvir; ombitasvir; paritaprevir; Viekira Pak; Ribavirin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ABT-450/r/ABT-267 and ABT-333, Plus RBV (Experimental): ABT-450/r/ABT-267 (150 mg/ 100 mg/ 25 mg once daily) and ABT-333 (250 mg twice daily), plus weight-based RBV (dosed 1,000 or 1,200 mg daily divided twice a day) for 12 weeks
  Interventions: Drug: ABT-450/r/ABT-267, ABT-333; Drug: Ribavirin
- ABT-450/r/ABT-267 and ABT-333, Plus Placebo RBV (Experimental): ABT-450/r/ABT-267 (150 mg/ 100 mg/ 25 mg once daily) and ABT-333 (250 mg twice daily) for 12 weeks plus placebo RBV (twice daily) for 12 weeks
  Interventions: Drug: ABT-450/r/ABT-267, ABT-333; Drug: Placebo for ribavirin

INTERVENTIONS:
Drug: ABT-450/r/ABT-267, ABT-333 — Tablet; ABT-450 coformulated with ritonavir and ABT-267, ABT-333 tablet
  Other Names: ABT-267 also known as ombitasvir; ABT-450 also known as paritaprevir; ABT-333 also known as dasabuvir; Viekira PAK
Drug: Ribavirin — Capsule
  Arms: ABT-450/r/ABT-267 and ABT-333, Plus RBV
Drug: Placebo for ribavirin — Capsule
  Arms: ABT-450/r/ABT-267 and ABT-333, Plus Placebo RBV

SUMMARY:
The purpose of this study is to evaluate the safety and antiviral activity of ABT-450/ritonavir/ABT-267 (ABT-450/r/ABT-267; ABT-450 also known as paritaprevir; ABT-267 also known as ombitasvir) and ABT-333 (also known as dasabuvir) with and without ribavirin (RBV) in patients with chronic hepatitis C virus genotype 1b (HCV GT1b) infection without cirrhosis.

DETAILED DESCRIPTION:
A randomized, double-blind, multicenter study to evaluate the safety and antiviral activity of the combination of ABT-450/ritonavir/ABT-267 (ABT-450/r/ABT-267) and ABT-333 with and without ribavirin (RBV) in treatment-naïve, noncirrhotic participants with chronic hepatitis C virus genotype 1b (HCV GT1b) infection.

ELIGIBILITY:
Inclusion Criteria:

* Females must be practicing specific forms of birth control on study treatment, or be post-menopausal for more than 2 years or surgically sterile
* Chronic hepatitis C, genotype 1b-infection (HCV RNA level greater than or equal to 10,000 IU/mL at screening)
* Subject has never received antiviral treatment for hepatitis C infection
* No evidence of liver cirrhosis

Exclusion Criteria:

* Significant liver disease with any cause other than HCV as the primary cause
* Positive hepatitis B surface antigen or anti-human immunodeficiency virus antibody
* Positive screen for drugs or alcohol
* Significant sensitivity to any drug
* Use of contraindicated medications within 2 weeks of dosing
* Abnormal laboratory tests

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 419 (Actual)
Dates: Start 2012-12; Primary Completion 2013-12 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dan Cohen, MD, Study Director — AbbVie

REFERENCES:
- [Background] Ferenci P, Bernstein D, Lalezari J, Cohen D, Luo Y, Cooper C, Tam E, Marinho RT, Tsai N, Nyberg A, Box TD, Younes Z, Enayati P, Green S, Baruch Y, Bhandari BR, Caruntu FA, Sepe T, Chulanov V, Janczewska E, Rizzardini G, Gervain J, Planas R, Moreno C, Hassanein T, Xie W, King M, Podsadecki T, Reddy KR; PEARL-III Study; PEARL-IV Study. ABT-450/r-ombitasvir and dasabuvir with or without ribavirin for HCV. N Engl J Med. 2014 May 22;370(21):1983-92. doi: 10.1056/NEJMoa1402338. Epub 2014 May 4. PMID 24795200
- [Derived] Feld JJ, Bernstein DE, Younes Z, Vlierberghe HV, Larsen L, Tatsch F, Ferenci P. Ribavirin dose management in HCV patients receiving ombitasvir/paritaprevir/ritonavir and dasabuvir with ribavirin. Liver Int. 2018 Sep;38(9):1571-1575. doi: 10.1111/liv.13708. Epub 2018 Mar 14. PMID 29377566
- See also: Related Info — http://rxabbvie.com

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | ABT-450/r/ABT-267 and ABT-333, Plus RBV | ABT-450/r/ABT-267 and ABT-333, Plus Placebo RBV
Started | 210 | 209
Completed | 208 | 207
Not Completed | 2 | 2
Not completed — Lost to Follow-up | 2 | 2

BASELINE CHARACTERISTICS:
Population: All randomized participants who received at least 1 dose of study drug
Groups:
- Total: Total of all reporting groups
Arm/Group | ABT-450/r/ABT-267 and ABT-333, Plus RBV | ABT-450/r/ABT-267 and ABT-333, Plus Placebo RBV | Total
Number analyzed (Participants) | 210 | 209 | 419
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.4 (11.94) | 49.2 (12.03) | 48.8 (11.98)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 104 | 123 | 227
  Male | 106 | 86 | 192

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Sustained Virologic Response 12 Weeks After Treatment; Noninferiority Analyses of Each Treatment Arm Compared to Historical Rate
Description: The percentage of participants with sustained virologic response (plasma Hepatitis C virus ribonucleic acid [HCV RNA] level less than the lower limit of quantitation [< LLOQ]) 12 weeks after the last dose of study drug. The LLOQ for the assay was 25 IU/mL.
  The primary efficacy endpoints were noninferiority of the percentage of participants who achieved sustained virologic response 12 weeks after treatment in each treatment arm (ABT-450/r/ABT-267 and ABT-333, plus either placebo RBV or RBV) compared with the historical control rate for noncirrhotic, treatment-naïve participants with HCV GT1b infection treated with telaprevir and peginterferon/RBV (pegIFN).
Time Frame: 12 weeks after last dose of study drug
Population: All randomized participants who received at least 1 dose of study drug (intent-to-treat [ITT] population); participants with missing data were counted as non-responders.
Measure: Number; unit: percentage of participants
Arm/Group | ABT-450/r/ABT-267 and ABT-333, Plus RBV | ABT-450/r/ABT-267 and ABT-333, Plus Placebo RBV
Number analyzed (Participants) | 210 | 209
percentage of participants | 99.5 | 100.0
Statistical Analysis 1: Comparison: ABT-450/r/ABT-267 and ABT-333, Plus Placebo RBV; For the primary efficacy endpoint of sustained virologic response at 12 weeks after treatment, based on a 2-sided significance level of 0.05 and an underlying rate of 92% or higher in each arm, a sample size of 200 participants per treatment arm provides >95% power to demonstrate noninferiority of each regimen to the historical rate for telaprevir plus pegIFN and RBV therapy (84%) (based on the normal approximation of a single binomial proportion in a one-sample test for superiority); Test type: Non-Inferiority or Equivalence — The noninferiority of the rate of sustained virologic response at 12 weeks after treatment for the ABT-450/r/ABT-267 and ABT-333, plus placebo RBV treatment group as compared with the historical rate for telaprevir plus pegIFN-RBV was analyzed; the lower confidence bound of the 2-sided 95% confidence interval (95% CI) for the percentage of participants with sustained virologic response at 12 weeks after treatment must exceed 73% to achieve noninferiority; Percentage of Participants = 100, 95% CI 2-sided [98.2 to 100.0] — 95% CI was calculated using the Wilson score method for the single proportion because the point estimate was 100%
Statistical Analysis 2: Comparison: ABT-450/r/ABT-267 and ABT-333, Plus RBV; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority or Equivalence — The noninferiority of the rate of sustained virologic response at 12 weeks after treatment for the ABT-450/r/ABT-267 and ABT-333, plus RBV treatment group as compared with the historical rate for telaprevir plus pegIFN-RBV was analyzed; the lower confidence bound of the 2-sided 95% CI for the percentage of participants with sustained virologic response at 12 weeks after treatment must exceed 73% to achieve noninferiority; Percentage of Participants = 99.5, 95% CI 2-sided [98.6 to 100.0] — 95% CI was calculated using the normal approximation to the binomial distribution

2. Secondary Outcome: Percentage of Participants With Sustained Virologic Response 12 Weeks After Treatment; Noninferiority Analysis of ABT-450/r/ABT-267 and ABT-333, Plus Placebo RBV Compared With ABT-450/r/ABT-267 and ABT-333, Plus RBV
Description: The percentage of participants with sustained virologic response (plasma Hepatitis C virus ribonucleic acid [HCV RNA] level less than the lower limit of quantitation [< LLOQ]) 12 weeks after the last dose of study drug.
  The secondary endpoint was the noninferiority of the percentage of participants who achieved sustained virologic response 12 weeks after treatment who received ABT-450/r/ABT-267 and ABT-333, plus placebo RBV compared with those who received ABT-450/r/ABT-267 and ABT-333, plus RBV.
Time Frame: 12 weeks after last dose of study drug
Population: All randomized participants who received at least 1 dose of study drug (ITT population); participants with missing data were counted as non-responders.
Measure: Number; unit: percentage of participants
Arm/Group | ABT-450/r/ABT-267 and ABT-333, Plus RBV | ABT-450/r/ABT-267 and ABT-333, Plus Placebo RBV
Number analyzed (Participants) | 210 | 209
percentage of participants | 99.5 | 100
Statistical Analysis 1: Comparison: ABT-450/r/ABT-267 and ABT-333, Plus RBV vs ABT-450/r/ABT-267 and ABT-333, Plus Placebo RBV; For the secondary efficacy endpoint of sustained virologic response at 12 weeks after treatment, based on a -10% margin, a 2-sided significance level of 0.05 and an underlying rate of 92% or higher in each arm, a sample size of 200 participants per arm provides >95% power to demonstrate noninferiority of ABT-450/r/ABT-267 and ABT-333, plus Placebo RBV compared with ABT-450/r/ABT-267 and ABT-333, plus RBV (normal approximation of a single binomial proportion in a 1-sample test for superiority); Test type: Non-Inferiority or Equivalence — Noninferiority of the rate of sustained virologic response at 12 weeks after treatment for the ABT-450/r/ABT-267 and ABT-333, plus placebo RBV treatment group as compared with the ABT-450/r/ABT-267 and ABT-333, plus RBV treatment group was analyzed using a noninferiority margin of -10.5%. The lower confidence bound of the 2-sided 95% CI for the difference in percentage of participants with sustained virologic response at 12 weeks after treatment must exceed -10.5% to achieve noninferiority; Difference in Percentage of Participants = 0.5, 95% CI 2-sided [-0.5 to 1.4] — 95% CI was calculated using the normal approximation to the binomial distribution

3. Secondary Outcome: Percentage of Participants With Hemoglobin Decrease to Below the Lower Limit of Normal (LLN) At End of Treatment
Description: The percentage of participants with a decrease in hemoglobin from greater than or equal to the lower limit of normal (≥ LLN) at baseline to < LLN at the end of treatment.
Time Frame: Baseline (Day 1) and Week 12 (End of Treatment)
Population: All randomized participants who received at least 1 dose of study drug (ITT population) and had hemoglobin ≥ LLN reference range at baseline.
Measure: Number; unit: percentage of participants
Arm/Group | ABT-450/r/ABT-267 and ABT-333, Plus RBV | ABT-450/r/ABT-267 and ABT-333, Plus Placebo RBV
Number analyzed (Participants) | 207 | 205
percentage of participants | 51.2 | 3.4
Statistical Analysis 1: Comparison: ABT-450/r/ABT-267 and ABT-333, Plus RBV vs ABT-450/r/ABT-267 and ABT-333, Plus Placebo RBV; Test type: Superiority or Other; p < 0.001, Fisher Exact

4. Secondary Outcome: Percentage of Participants With Sustained Virologic Response 12 Weeks After Treatment; Superiority Analyses of Each Treatment Arm Compared to Historical Rate
Description: The percentage of participants with sustained virologic response (plasma HCV RNA less than the lower limit of quantitation [< LLOQ]) 12 weeks after the last dose of study drug.
  The secondary efficacy endpoints were superiority of the percentage of participants who achieved sustained virologic response 12 weeks after treatment in each treatment arm (ABT-450/r/ABT-267 and ABT-333, plus either placebo RBV or RBV) compared with the historical control rate for noncirrhotic, treatment-naïve participants with HCV GT1b treated with telaprevir and pegIFN/RBV.
Time Frame: 12 weeks after last dose of study drug
Population: as for outcome 2
Measure: Number; unit: percentage of particpants
Arm/Group | ABT-450/r/ABT-267 and ABT-333, Plus RBV | ABT-450/r/ABT-267 and ABT-333, Plus Placebo RBV
Number analyzed (Participants) | 210 | 209
percentage of particpants | 99.5 | 100
Statistical Analysis 1: Comparison: ABT-450/r/ABT-267 and ABT-333, Plus Placebo RBV; For the secondary efficacy endpoint of sustained virologic response at 12 weeks after treatment, based on a 2-sided significance level of 0.05 and an underlying rate of 92% or higher in each arm, a sample size of 200 participants per treatment arm provides >90% power to demonstrate superiority of each regimen to the historical rate for telaprevir plus pegIFN and RBV therapy (84%) (based on the normal approximation of a single binomial proportion in a one-sample test for superiority); Test type: Superiority or Other; Percentage of Participants = 100, 95% CI 2-sided [98.2 to 100.0] — 95% CI calculated using the Wilson score method for the single proportion; the lower confidence bound for the percentage of participants with sustained virologic response at 12 weeks after treatment must exceed 84% to achieve superiority
Statistical Analysis 2: Comparison: ABT-450/r/ABT-267 and ABT-333, Plus RBV; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; Percentage of Participants = 99.5, 95% CI 2-sided [98.6 to 100.0] — 95% CI calculated using the normal approximation to the binomial distribution; the lower confidence bound for the percentage of participants with sustained virologic response at 12 weeks after treatment must exceed 84% to achieve superiority

5. Secondary Outcome: Percentage of Participants With Virologic Failure During Treatment
Description: Virologic failure during treatment was defined as rebound (confirmed HCV RNA greater than or equal to the lower limit of quantitation [≥ LLOQ] after HCV RNA < LLOQ during treatment, or confirmed increase from the lowest value post baseline in HCV RNA [2 consecutive HCV RNA measurements > 1 log10 IU/mL above the lowest value post baseline] at any time point during treatment), or failure to suppress (HCV RNA ≥ LLOQ persistently during treatment with at least 6 weeks [≥ 36 days] of treatment).
Time Frame: Baseline (Day 1), and Treatment Weeks 1, 2, 4, 6, 8, 10, and 12
Population: All randomized participants who received at least 1 dose of study drug (ITT population).
Measure: Number; unit: percentage of participants
Arm/Group | ABT-450/r/ABT-267 and ABT-333, Plus RBV | ABT-450/r/ABT-267 and ABT-333, Plus Placebo RBV
Number analyzed (Participants) | 210 | 209
percentage of participants
  Rebound | 0.5 | 0
  Failure to suppress | 0 | 0

6. Secondary Outcome: Percentage of Participants With Virologic Relapse After Treatment
Description: Participants who completed treatment with plasma HCV RNA less than the lower limit of quantification (<LLOQ) at the end of treatment were considered to have virologic relapse if they had confirmed HCV RNA ≥ LLOQ during the post-treatment period.
Time Frame: Between End of Treatment (Week 12) and Post-treatment (up to Week 12 Post-treatment)
Population: All randomized participants who received at least 1 dose of study drug (ITT population) with HCV RNA < LLOQ at the final treatment visit and completed treatment.
Measure: Number; unit: percentage of participants
Arm/Group | ABT-450/r/ABT-267 and ABT-333, Plus RBV | ABT-450/r/ABT-267 and ABT-333, Plus Placebo RBV
Number analyzed (Participants) | 208 | 207
percentage of participants | 0 | 0

ADVERSE EVENTS:
Time Frame: AEs were collected from the time of study drug administration to 30 days after last dose of study drug (16 weeks); SAEs were also collected from the time that informed consent was obtained until the end of participation in the study (up to 65 weeks)
Arm/Group | ABT-450/r/ABT-267 and ABT-333, Plus RBV | ABT-450/r/ABT-267 and ABT-333, Plus Placebo RBV
Serious Adverse Events (participants affected / at risk) | 4/210 | 4/209
Other Adverse Events (participants affected / at risk) | 133/210 | 97/209
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ABT-450/r/ABT-267 and ABT-333, Plus RBV (N=210) | ABT-450/r/ABT-267 and ABT-333, Plus Placebo RBV (N=209)
ATRIAL FIBRILLATION (Cardiac disorders) | 1 | 0
CORONARY ARTERY DISEASE (Cardiac disorders) | 1 | 0
ARTHRITIS (Musculoskeletal and connective tissue disorders) | 0 | 1
MYALGIA (Musculoskeletal and connective tissue disorders) | 0 | 1
INTRADUCTAL PROLIFERATIVE BREAST LESION (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
NEPHROLITHIASIS (Renal and urinary disorders) | 1 | 0
EPIDIDYMITIS (Reproductive system and breast disorders) | 1 | 0
UTERINE POLYP (Reproductive system and breast disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | ABT-450/r/ABT-267 and ABT-333, Plus RBV (N=210) | ABT-450/r/ABT-267 and ABT-333, Plus Placebo RBV (N=209)
ANAEMIA (Blood and lymphatic system disorders) | 14 | 1
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 11 | 6
DIARRHOEA (Gastrointestinal disorders) | 9 | 13
DYSPEPSIA (Gastrointestinal disorders) | 14 | 9
NAUSEA (Gastrointestinal disorders) | 23 | 9
ASTHENIA (General disorders) | 22 | 12
FATIGUE (General disorders) | 45 | 49
HEADACHE (Nervous system disorders) | 51 | 49
INSOMNIA (Psychiatric disorders) | 19 | 7
COUGH (Respiratory, thoracic and mediastinal disorders) | 19 | 5
PRURITUS (Skin and subcutaneous tissue disorders) | 25 | 11
RASH (Skin and subcutaneous tissue disorders) | 12 | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.